CLINICAL TRIAL: NCT04724252
Title: Gabapentin to Reduce Opioid Use Postoperatively (GROUP) in Children
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1571754
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pain, Postoperative
Keywords: thoracic surgery; cardiac surgery via a sternotomy or thoracotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Children meeting criteria will be randomized in a 1:1 ratio using 4 blocked randomization to either gabapentin or placebo (in addition to standard of care pain control treatment):
Who Masked: Participant, Investigator
Masking Description: This study is a double-blind, placebo controlled, randomized study. Physician and families will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Gabapentin Treatment (Active Comparator): Given at a dose of 10mg/kg (max 600mg) perioperatively (immediately prior to surgery) followed by 3mg/kg/dose TID with first dose to be given starting at 8 hours post perioperative dose.
  Interventions: Drug: Gabapentin
- Control Group (Placebo Comparator): Given placebo which coincides with the active treatment group
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Determine if the peri and post operative use of gabapentin in children reduces the need for narcotics after surgery.
  Arms: Gabapentin Treatment
Other: Placebo — Control Arm
  Arms: Control Group

SUMMARY:
The primary objective of this study is to determine if the peri and post operative use of gabapentin in children reduces the need for narcotics after thoracic surgery.

We hypothesize that patients who are given gabapentin will need fewer morphine equivalents postoperatively than those who were not given gabapentin

DETAILED DESCRIPTION:
This study is a double-blind, placebo controlled, randomized study to explore the effects of gabapentin peri and post operatively. Physician and families will be blinded to the treatment.

60 subjects will be randomized in a 1:1 ratio to either:

* Gabapentin treatment group
* Placebo - control group

We aim to understand the impact that gabapentin use peri and post operatively has on:

1. opioid use based of IV morphine
2. pain scores
3. opioid related complications such as withdrawal
4. effects on the level of sedation
5. Possible adverse effects associated with use of gabapentin
6. Time to extubating

The duration of an individual subject's participation in the study will be 7 days or until the patient is discharged from UC Davis Hospital, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age newborn to < 18 years.
2. Gestational age to be minimum 38 weeks.
3. Undergo cardiac surgery via a sternotomy or thoracotomy. OR Any Thoracic Surgery OR Planned noncardiac surgery via a thoracotomy or Video Assisted Thoracotomy (VATS).
4. Surgery will result in an inpatient stay of at least 48 hours.

Exclusion Criteria:

1. Use of opioids within 30 days prior to study entry.
2. Renal Failure as defined by RIFLE Criteria.
3. History of seizures requiring active treatment.
4. History of chronic pain treated medically.
5. Diagnosis of Autism.
6. Unable to tolerate enteral medications.
7. Hematology/Oncology patients.
8. Parents/legal guardians unable to consent.
9. Participation in another clinical study presently or within the last 30 days
10. Pregnancy
11. Prisoners
12. Patient undergoing nuss procedure with cryoablation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amount of pain medication needed. | 7 days post-operative or until discharge, whichever came first
  Amount of pain medication needed after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-gabapentin-to-reduce-opioid-use-after-surgery-in-children-the-group-study-210128/